CLINICAL TRIAL: NCT02679261
Title: Evaluating the Effectiveness of Atorvastatin on the Progression of Aortic Dilatation and Valvular Degeneration in Patients With Bicuspid Aortic Valve (BICATOR)
Brief Title: Evaluating the Effectiveness of Atorvastatin on the Progression of Aortic Dilatation and Valvular Degeneration in Patients With Bicuspid Aortic Valve
Acronym: BICATOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BICATOR
Record Dates: First submitted 2016-01-19; First posted 2016-02-10 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Bicuspid Aortic Valve
Keywords: Aortic dilation; Statins; Aortic degeneration
MeSH Terms: conditions — Bicuspid Aortic Valve Disease | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): Oral administration Atorvastatin 20 mg per day
  Interventions: Drug: Atorvastatin
- Control (Placebo Comparator): Oral administration of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Oral administration atorvastatin 20 mg per day
  Arms: Atorvastatin
Drug: Placebo — Oral administration placebo
  Arms: Control

SUMMARY:
Bicuspid Aortic Valve (BAV) is the most common congenital heart disease affecting 1-2% of the population. The aortic dilation and aortic valve degeneration are common complications in patients with BAV. Statins have shown a reduction in the expression of metalloproteinases of the extracellular matrix observed in aortic aneurisms. Several retrospective studies have suggested the benefit of the statins to reduce aortic dilation in patients with BAV. Moreover, although statins did not show to be useful in the progression of aortic stenosis, different studies have suggested a higher profit when the valve affection is not severe. The objective of this study is to determine whether atorvastatin is effective at reducing the progression of aortic dilation in patients with BAV.

DETAILED DESCRIPTION:
BICATOR is a multicentre (8 centres), randomised, double-blind and placebo-controlled clinical trial aimed at evaluating the effect of atorvastatin in reducing progression of aortic dilation in patients with BAV. The primary outcome is to determine whether atorvastatin is effective in reducing aortic dilation in BAV and secondary outcome is to define if atorvastatin treatment slows the progression of aortic valve degeneration (valve calcification) in a 3 year follow-up period. 220 patients will be included (110 atorvastatin - 110 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old with BAV confirmed by transthoracic echocardiography (in case of doubts other techniques will be required: transesophageal echocardiography or CT to confirm diagnosis).
* Valve dysfunction only moderate: in case of aortic stenosis with average gradient < 30 mmHg and in case of aortic regurgitation a vena contracta < 7 mm or a jet with < 10 mm.
* Aortic valve not show severe calcification by transthoracic echocardiography.
* Ascending aortic diameter (Valsalva sinus or tubular ascending aorta) ≤ 50 mm.
* The patient must give the consent form signed.

Exclusion Criteria:

* Patients younger than 18.
* Patients with uncontrolled hypertension and a history or risk of diabetes mellitus.
* Patients who receive statins treatment or other lipid lowering drug or if they have indication to be treated according to the current clinical practice guidelines.
* Previous cardiac surgery or any surgery of other segments of the aorta.
* Previous aortic dissection and/or aortic coarctation.
* NYHA functional class III or IV.
* Presence or antecedent of liver failure (transaminase > 2 fold the superior limit of normal levels according to local laboratory), renal failure (creatinine clearance < 30ml/min or creatinine > 2.5mg/dl), myopathy or creatine kinase levels > 5 fold the superior limit of normality, or other gastrointestinal, hematologic or endocrine diseases or any other situation that according to the investigator criteria could affect the study treatment evaluation.
* Hypersensitivity, intolerance or contraindication to any component of the study drug or to the contrast used in CT.
* Pregnancy, breastfeeding or desire for pregnancy during the study period. A negative pregnancy test (negative gonadotropin) will be required in all fertile women to participate in the study.
* Participation in another drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Change of the diameter of ascending aorta by CT (Computed Tomography). | 3 years
  Determination of the progression of ascending aortic dilation assessed by measuring the change of the diameter of ascending aorta by CT (Computed Tomography).The change of the aortic diameter will be defined by the major difference between the measurements taken in the aortic root and ascending aorta in the initial and final study.

SECONDARY OUTCOMES:
Change of the final maximum diameter of the aortic root and the basal measured by CT. | 3 years
  Difference between the final maximum diameter of the aortic root and the basal measured by CT.
Change of the final maximum diameter of the tubular ascending aorta and the basal measured by CT. | 3 years
  Difference between the final maximum diameter of the tubular ascending aorta and the basal measured by CT.
Change of the final area of the aortic root and the basal measured by CT. | 3 years
  Difference between the final area of the aortic root and the basal measured by CT.
Change of the the final area of ascending aorta and the basal measured by CT. | 3 years
  Difference between the final area of ascending aorta and the basal measured by CT.
Change of the valve Agatston final score and the basal assessed by CT. | 3 years
  Difference between the valve Agatston final score and the basal assessed by CT.
Change of the final planimetry area of the aortic valve and the basal measured by CT. | 3 years
  Difference between the final planimetry area of the aortic valve and the basal measured by CT.
Change of the transvalvular pressure gradient of the aortic valve | 3 years
  Difference of transvalvular pressure gradient of the aortic valve
Change of aortic regurgitation jet width basal and final. | 3 years
  Difference of aortic regurgitation jet width basal and final.
Change of the maximum aortic velocity | 3 years
  Change of the maximum aortic velocity
Change of aortic valve area | 3 years
  Change of aortic valve area by continuity equation basal and final
Ocurrence of Serious Adverse Clinical Events leading to hospitalization and death | 3 years
  Serious Adverse Clinical Events: Aortic dissection, aortic rupture or need for aortic surgery, cardiovascular death, death of any cause. Combined endpoint of death, aortic dissection or need for aortic or valve surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Evangelista-Masip, MD, PhD, Professor, Principal Investigator — Hospital Universitari Vall d'Hebron, Vall d'Hebron Institut de Recerca
Locations (10):
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Clínico Universitario de Valladolid, Valladolid

REFERENCES:
- [Background] Crisby M, Nordin-Fredriksson G, Shah PK, Yano J, Zhu J, Nilsson J. Pravastatin treatment increases collagen content and decreases lipid content, inflammation, metalloproteinases, and cell death in human carotid plaques: implications for plaque stabilization. Circulation. 2001 Feb 20;103(7):926-33. doi: 10.1161/01.cir.103.7.926. PMID 11181465
- [Background] Schouten O, van Laanen JH, Boersma E, Vidakovic R, Feringa HH, Dunkelgrun M, Bax JJ, Koning J, van Urk H, Poldermans D. Statins are associated with a reduced infrarenal abdominal aortic aneurysm growth. Eur J Vasc Endovasc Surg. 2006 Jul;32(1):21-6. doi: 10.1016/j.ejvs.2005.12.024. Epub 2006 Mar 6. PMID 16520071
- [Background] Sukhija R, Aronow WS, Sandhu R, Kakar P, Babu S. Mortality and size of abdominal aortic aneurysm at long-term follow-up of patients not treated surgically and treated with and without statins. Am J Cardiol. 2006 Jan 15;97(2):279-80. doi: 10.1016/j.amjcard.2005.08.033. Epub 2005 Nov 21. PMID 16442379
- [Background] McLoughlin D, McGuinness J, Byrne J, Terzo E, Huuskonen V, McAllister H, Black A, Kearney S, Kay E, Hill AD, Dietz HC, Redmond JM. Pravastatin reduces Marfan aortic dilation. Circulation. 2011 Sep 13;124(11 Suppl):S168-73. doi: 10.1161/CIRCULATIONAHA.110.012187. PMID 21911808
- [Background] Jovin IS, Duggal M, Ebisu K, Paek H, Oprea AD, Tranquilli M, Rizzo J, Memet R, Feldman M, Dziura J, Brandt CA, Elefteriades JA. Comparison of the effect on long-term outcomes in patients with thoracic aortic aneurysms of taking versus not taking a statin drug. Am J Cardiol. 2012 Apr 1;109(7):1050-4. doi: 10.1016/j.amjcard.2011.11.038. Epub 2012 Jan 3. PMID 22221941
- [Background] Stein LH, Berger J, Tranquilli M, Elefteraides JA. Effect of statin drugs on thoracic aortic aneurysms. Am J Cardiol. 2013 Oct 15;112(8):1240-5. doi: 10.1016/j.amjcard.2013.05.081. PMID 24079445
- [Background] Goel SS, Tuzcu EM, Agarwal S, Aksoy O, Krishnaswamy A, Griffin BP, Svensson LG, Kapadia SR. Comparison of ascending aortic size in patients with severe bicuspid aortic valve stenosis treated with versus without a statin drug. Am J Cardiol. 2011 Nov 15;108(10):1458-62. doi: 10.1016/j.amjcard.2011.06.071. PMID 22040719
- [Background] Cowell SJ, Newby DE, Prescott RJ, Bloomfield P, Reid J, Northridge DB, Boon NA; Scottish Aortic Stenosis and Lipid Lowering Trial, Impact on Regression (SALTIRE) Investigators. A randomized trial of intensive lipid-lowering therapy in calcific aortic stenosis. N Engl J Med. 2005 Jun 9;352(23):2389-97. doi: 10.1056/NEJMoa043876. PMID 15944423
- [Background] Dichtl W, Alber HF, Feuchtner GM, Hintringer F, Reinthaler M, Bartel T, Sussenbacher A, Grander W, Ulmer H, Pachinger O, Muller S. Prognosis and risk factors in patients with asymptomatic aortic stenosis and their modulation by atorvastatin (20 mg). Am J Cardiol. 2008 Sep 15;102(6):743-8. doi: 10.1016/j.amjcard.2008.04.060. Epub 2008 Jul 2. PMID 18774000
- [Background] Moura LM, Ramos SF, Zamorano JL, Barros IM, Azevedo LF, Rocha-Goncalves F, Rajamannan NM. Rosuvastatin affecting aortic valve endothelium to slow the progression of aortic stenosis. J Am Coll Cardiol. 2007 Feb 6;49(5):554-61. doi: 10.1016/j.jacc.2006.07.072. Epub 2007 Jan 22. PMID 17276178
- [Background] Chan KL, Teo K, Dumesnil JG, Ni A, Tam J; ASTRONOMER Investigators. Effect of Lipid lowering with rosuvastatin on progression of aortic stenosis: results of the aortic stenosis progression observation: measuring effects of rosuvastatin (ASTRONOMER) trial. Circulation. 2010 Jan 19;121(2):306-14. doi: 10.1161/CIRCULATIONAHA.109.900027. Epub 2010 Jan 4. PMID 20048204
- [Background] Rossebo AB, Pedersen TR, Boman K, Brudi P, Chambers JB, Egstrup K, Gerdts E, Gohlke-Barwolf C, Holme I, Kesaniemi YA, Malbecq W, Nienaber CA, Ray S, Skjaerpe T, Wachtell K, Willenheimer R; SEAS Investigators. Intensive lipid lowering with simvastatin and ezetimibe in aortic stenosis. N Engl J Med. 2008 Sep 25;359(13):1343-56. doi: 10.1056/NEJMoa0804602. Epub 2008 Sep 2. PMID 18765433
- [Background] Antonini-Canterin F, Hirsu M, Popescu BA, Leiballi E, Piazza R, Pavan D, Ginghina C, Nicolosi GL. Stage-related effect of statin treatment on the progression of aortic valve sclerosis and stenosis. Am J Cardiol. 2008 Sep 15;102(6):738-42. doi: 10.1016/j.amjcard.2008.04.056. Epub 2008 Jun 26. PMID 18773999
- [Derived] Evangelista A, Galian-Gay L, Guala A, Teixido-Tura G, Calvo-Iglesias F, Sevilla T, Bermejo J, Mendez I, Sanchez V, Robledo Carmona JM, Alegret JM, Ferrer-Sistach E, Saura D, Ruiz-Munoz A, Dux-Santoy L, Carmona MA, Huguet M, Cuellar-Calabria H, Sao-Aviles A, Ferreira-Gonzalez I, Rodriguez-Palomares JF. Atorvastatin Effect on Aortic Dilatation and Valvular Calcification Progression in Bicuspid Aortic Valve (BICATOR): A Randomized Clinical Trial. Circulation. 2024 Jun 18;149(25):1938-1948. doi: 10.1161/CIRCULATIONAHA.123.067537. Epub 2024 May 28. PMID 38804148